CLINICAL TRIAL: NCT01855568
Title: Comparison of Two-dose and Single-dose Methotrexate Protocol for Ectopic Pregnancy: a Randomized Controlled Trial
Brief Title: Methotrexate Treatment for Ectopic Pregnancy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CHA University (Other)
Responsible Party: Principal Investigator, Taejong Song, Professor, CHA University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KNC13-006
Record Dates: First submitted 2013-05-10; First posted 2013-05-16 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2016-01

CONDITIONS: Ectopic Pregnancy
MeSH Terms: conditions — Pregnancy, Ectopic | interventions — Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single-dose methotrexate protocol (Experimental): Participants in the "single-dose protocol" group received intramuscular methotrexate at single dose of 50 mg/m2 on day 0 (the initial day of treatment). The β-hCG levels were then measured on day 4 and 7. If there was at least 15% β-hCG drop between day 4 and 7, the treatment was deemed successful and the participants were then followed with weekly β-hCG measurements until the results was negative. If a 15% drop on day 4 and 7 did not occur, a second dose was administrated on day 7 and β-hCG levels were then measured on day 11 and 14. Participants were referred for surgical treatment if β-hCG levels fell <15% between day 11 and 14.
  Interventions: Procedure: Single-dose Methotrexate
- Two-dose methotrexate protocol (Experimental): Participants in the "two-dose protocol" group received intramuscular methotrexate twice at dose of 50 mg/m2 on day 0 and 4. A third dose of methotrexate was given on day 7 if β-hCG levels did not fall 15% between day 4 and 7 after two-dosing. A fourth dose was administered on day 11 if β-hCG levels fell <15% between day 7 and 11. Then, a final β-hCG level was checked on day 14. If a 15% drop was not seen, the medical treatment was deemed refractory and the patients were referred for surgical treatment.
  Interventions: Procedure: Two-dose methotrexate protocol

INTERVENTIONS:
Procedure: Single-dose Methotrexate — Participants in the "single-dose protocol" group received intramuscular methotrexate at single dose of 50 mg/m2 on day 0 (the initial day of treatment). The β-hCG levels were then measured on day 4 and 7. If there was at least 15% β-hCG drop between day 4 and 7, the treatment was deemed successful and the participants were then followed with weekly β-hCG measurements until the results was negative. If a 15% drop on day 4 and 7 did not occur, a second dose was administrated on day 7 and β-hCG levels were then measured on day 11 and 14. Participants were referred for surgical treatment if β-hCG levels fell <15% between day 11 and 14.
  Arms: Single-dose methotrexate protocol
Procedure: Two-dose methotrexate protocol — Participants in the "two-dose protocol" group received intramuscular methotrexate twice at dose of 50 mg/m2 on day 0 and 4. A third dose of methotrexate was given on day 7 if β-hCG levels did not fall 15% between day 4 and 7 after two-dosing. A fourth dose was administered on day 11 if β-hCG levels fell <15% between day 7 and 11. Then, a final β-hCG level was checked on day 14. If a 15% drop was not seen, the medical treatment was deemed refractory and the patients were referred for surgical treatment.
  Arms: Two-dose methotrexate protocol

SUMMARY:
Ectopic pregnancy is an important cause of maternal morbidity and occasionally mortality. Deaths associated with ectopic pregnancy have declined, though approximately 75% of deaths in the first trimester and 9-13% of all pregnancy-related deaths are associated ectopic pregnancy. The main stays of management for ectopic pregnancy were surgery and medical treatment. Medical management with systemic methotrexate administration avoids the inherent morbidity of anesthesia and surgery is cost-effective, and also offers success rates comparable to surgical management, with no loss in future potential fertility.

However, although medical management using methotrexate is used commonly, there is no solid consensus regarding dose protocol. Currently, there are three methotrexate protocols for the treatment of an ectopic pregnancy, "multi-dose", "single-dose", or "two-dose". Among them, the multi-dose protocol includes the administration of 4 methotrexate doses alternating with leucovorin (rescue regimen). As a result of the multiple dosing of methotrexate, side effects are more common. In contrast, the advantages of the single-dose protocol include elimination of a rescue regimen, lower incidence of adverse effects, and better compliance. However, the single-dose protocol was found to be associated with a considerably lower success rate as compared with the multi-dose protocol (88% versus 93%) in a recent meta-analysis. The two-dose protocol, which it balances efficacy and safety/convenience, was described as a cross between the multi-dose and single-dose protocols.

However, there were a few studies comparing between single-dose and two-dose protocol. The purpose of this prospective randomized trial was to compared the success rates of single-dose and two-dose methotrexate protocol for the treatment of tubal ectopic pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* tubal pregnancy
* tubal pregnancy except interstitial pregnancy
* a pretreatment β-hCG level <15000 mIU/mL
* a gestational sac with a largest diameter <4 cm
* hemodynamically stable status
* agreement to methotrexate treatment and follow up

Exclusion Criteria:

* heterotrophic pregnancy
* a presence of embryonic cardiac motion
* clinically or sonographically suspected tubal rupture
* laboratory tests showing possible deleterious effects of methotrexate treatment on organ functions

Ages: 19 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2013-05; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
treatment success | Up to 8 weeks (normal recovery time after treatment)
  Participants in both groups were considered a treatment success if β-hCG levels resolved to <5 mIU/mL without surgical intervention. The cases of participants who underwent surgical intervention were considered to have had treatment failure.

CONTACTS AND LOCATIONS:
Overall Officials: Taejong Song, M.D., Principal Investigator — CHA Gangnam Medical Center, Seoul, Republic of Korea
Locations (1):
- CHA Gangnam Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Song T, Kim MK, Kim ML, Jung YW, Yun BS, Seong SJ. Single-dose versus two-dose administration of methotrexate for the treatment of ectopic pregnancy: a randomized controlled trial. Hum Reprod. 2016 Feb;31(2):332-8. doi: 10.1093/humrep/dev312. Epub 2015 Dec 23. PMID 26701971